CLINICAL TRIAL: NCT02205489
Title: Single Arm Study To Assess Comprehensive Infusion Guidance For The Management Of The Infusion- Associated Reactions (IARs) In Relapsing-Remitting Multiple Sclerosis (RRMS) Patients Treated With LEMTRADA
Brief Title: Management Of The Infusion-Associated Reactions In RRMS Patients Treated With LEMTRADA
Acronym: EMERALD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS13650; 2014-000092-62; U1111-1153-3922 (Other: UTN)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Alemtuzumab; Cetirizine; Ranitidine; Methylprednisolone; Acyclovir; Esomeprazole; Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GZ402673 LEMTRADA (Experimental): First course: Intravenous infusion for 5 consecutive days. Second course (will occur 12 months after the first course of treatment): Intravenous infusion for 3 consecutive days.
  Interventions: Drug: Alemtuzumab GZ402673; Drug: cetirizine; Drug: ranitidine; Drug: methylprednisolone; Drug: aciclovir; Drug: esomeprazole; Drug: ibuprofen; Drug: paracetamol

INTERVENTIONS:
Drug: Alemtuzumab GZ402673 — Pharmaceutical form:concentration for solution Route of administration: intravenous infusion
  Other Names: Lemtrada
Drug: cetirizine — Pharmaceutical form:tablet Route of administration: oral
Drug: ranitidine — Pharmaceutical form:tablet Route of administration: oral
Drug: methylprednisolone — Pharmaceutical form:tablet Route of administration: oral
Drug: methylprednisolone — Pharmaceutical form:solution Route of administration: intravenous
Drug: aciclovir — Pharmaceutical form:tablet Route of administration: oral
Drug: esomeprazole — Pharmaceutical form:tablet Route of administration: oral
Drug: ibuprofen — Pharmaceutical form:tablet Route of administration: oral
Drug: paracetamol — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To assess the distribution of IARs by severity grade when LEMTRADA is administered to RRMS patients who will be medicated according to specified algorithm designed to manage infusion associated reactions.

DETAILED DESCRIPTION:
The total duration of participation in the study per patient is approximately 13.5 months.

After the end of the second course of LEMTRADA treatment, patients will be followed by their physician in a regular healthcare setting until 48 months safety monitoring period is completed.

ELIGIBILITY:
Inclusion criteria:

* Adult RRMS patients who will be initiating treatment with Lemtrada according to local approved label.
* Signed written informed consent.

Exclusion criteria:

* Previously treated with LEMTRADA.
* Contraindications to LEMTRADA according to the labeling in the country.
* Any known contraindications to the symptomatic therapy used in the infusion management guidance based on their local approved label.
* Currently participating in another investigational interventional study.
* Any technical/administrative reason that makes it impossible to enroll the patient in the study.
* Patient is the Investigator or any Sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Patient who has withdrawn consent before enrollment (starting from signed informed consent form).
* Despite screening of the patient, enrolment is stopped at the study level.
* Woman of childbearing potential not protected by highly-effective method(s) of birth control (as defined in a local protocol amendment in case of specific local requirement) and/or who are unwilling or unable to be tested for pregnancy.
* Pregnancy (defined as positive beta human chorionic gonadotropin (β-HCG) blood test), breast feeding.
* Known infection with latent tuberculosis or active tuberculosis.
* Known infection with Hepatitis B, Hepatitis C.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of IARs that are graded mild according to the Common Toxicity Criteria (CTC). An IAR is any adverse event occurring during or within 24 hours of LEMTRADA infusion. | up to 30 days in the first treatment course and the second treatment course, respectively
Proportion of IARs | up to 30 days in the first treatment course and the second treatment course, respectively
Proportion and type of serious IARs | up to 30 days in the first treatment course and the second treatment course, respectively
Proportion by type (as defined by clinical symptoms) | up to 30 days in the first treatment course and the second treatment course, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- Belgium (2):
  - Investigational Site Number 056002, Bruges
  - Investigational Site Number 056001, Brussels
- France (10):
  - Investigational Site Number 250009, Dijon
  - Investigational Site Number 250005, Lille
  - Investigational Site Number 250001, Lyon Bron
  - Investigational Site Number 250006, Nancy
  - Investigational Site Number 250010, Nantes
  - Investigational Site Number 250007, Nîmes
  - Investigational Site Number 250008, Paris
  - Investigational Site Number 250004, Rennes
  - Investigational Site Number 250003, Strasbourg
  - Investigational Site Number 250002, Toulouse
- Netherlands (2):
  - Investigational Site Number 528001, Breda
  - Investigational Site Number 528002, Rotterdam
- Spain (6):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724005, Bilbao
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724006, Málaga
  - Investigational Site Number 724003, Seville
  - Investigational Site Number 724004, Valencia